CLINICAL TRIAL: NCT01332630
Title: A Phase 2 Open-Label Study of TPI 287 in Patients With Breast Cancer Metastatic to the Brain
Brief Title: TPI 287 in Breast Cancer Metastatic to the Brain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cortice Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0198; NCI-2011-00929 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Results first posted 2018-07-10 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Brain metastases; TPI 287; Computed Tomography; CT; Magnetic Resonance Imaging; MRI
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — TPI-287; Dexamethasone; Calcium Dobesilate; Diphenhydramine; Ranitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TPI 287 (Experimental): TPI 287 administered at 160 mg/m2 by vein on Day 1 and repeated every three weeks. Day 1 of each subsequent cycle is equivalent of day 22 of the previous cycle; pre TPI 287: Dexamethasone 6 mg by mouth at 12 hours and 6 hours prior to treatment. As alternative and based on the treating physician discretion, Dexamethasone 10 mgby vein may be given 30-60 minutes prior to treatment with TPI 287, Benadryl 12.5-25 mg IV push over 30-60 minutes, and Ranitidine 1mg/kg IV over 30-60 minutes.
  Interventions: Drug: TPI 287; Drug: Dexamethasone; Drug: Benadryl; Drug: Ranitidine

INTERVENTIONS:
Drug: TPI 287 — Starting dose Phase I: 160 mg/m2 by vein over 60 minutes on Days 1, 8, and 15 of every 28 day cycle.
  Starting Dose Phase II: Maximum tolerated dose from Phase I.
Drug: Dexamethasone — 6 mg by mouth at 12 hours and 6 hours prior to treatment. As alternative and based on the treating physician discretion, dexamethasone 10 mg by vein may be given 30-60 minutes prior to treatment with TPI 287.
  Other Names: Decadron
Drug: Benadryl — 12.5-25 mg intravenous (IV) push 30-60 minutes prior
  Other Names: Diphenhydramine
Drug: Ranitidine — As H2 blocker 1mg/kg IV 30-60 minutes prior
  Other Names: Zantac; Ranitidine hydrochloride

SUMMARY:
The goal of the first part of this clinical research study is to find the highest tolerable dose of TPI-287 in patients with breast cancer that has spread to the brain.

The goal of the second part of this study is to learn if TPI-287 can control breast cancer that has spread to the brain. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

TPI-287 is designed to prevent cancer cells from dividing, which may slow and/or stop the growth of cancer cell.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive, TPI 287 by vein over 60 minutes on Day 1 of every 21 day cycle.

Before you receive the study drug, you will receive dexamethasone by mouth, Benadryl (diphenhydramine HCL) by vein over 30-60 minutes, and ranitidine over 30-60 minutes to help prevent a potential serious allergic reaction.

Study Visits:

At all study visits, you will be asked about any side effects you may be having and about any other drugs you may be taking.

On Days 1, 8, and 15 of Cycle 1, blood (about 2-3 teaspoons) will be drawn for routine tests. If you are taking coumadin, blood (about 1-2 teaspoons) will be drawn to check how well your blood clots.

On Day 1 of Cycle 1, your performance status will be recorded and your vital signs will be measured.

Within 7 days of Day 1 of Cycles 2 and beyond:

* Blood (about 2-3 tablespoons) will be drawn for routine tests. If you are taking coumadin, blood (about 1-2 teaspoons) will be drawn to check how well your blood clots.
* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will have a neurological exam.

Every 6 weeks (that is, before each odd-numbered cycle):

* You may have CT scans or MRI scans of the chest, abdomen, and pelvis to check the status of the disease.
* You will have a MRI of your brain. The MRI will require a catheter to be inserted into one of your veins in order to inject the MRI contrast agent.

The study doctor and staff will review your imaging scans to check what stage of disease the tumors inside and/or outside your brain are.

Length of Study:

You may continue to receive TPI 287 for as long as the doctor thinks it is in your best interest. You will no longer be able to receive TPI 287 if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after you have completed the end-of-treatment and follow-up visits.

End-of Treatment Visit:

About 4 weeks after you stop taking TPI 287:

* You will have a physical exam, including measurement of your vital signs.
* You will have a neurological exam.
* Your performance status will be measured.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* You will have a CT and/or MRI to check the status of the disease. This may include a brain MRI. If your doctor thinks it is needed, you will have a bone scan.
* You will be asked about any side effects you may have had any drugs you may be taking.

Follow-Up Visits:

Once you are off-study, you will be contacted either in the clinic or by phone every 3 months for up to 1 year after you enrolled on the study to check on the status of your health. If you are called, it will take less than 5 minutes.

This is an investigational study. TPI 287 is not FDA approved or commercially available. At this time, TPI 287 is being used in research only.

Up to 69 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically proven breast cancer with metastatic disease to the brain.
2. Patients must have measurable disease on MRI that has progressed after prior therapy. PD will be defined as a>/= 25% increase in the sum of the products of greatest perpendicular diameters of all measurable disease over the smallest sum observed (since treatment started) on Gd-MRI, the appearance of new lesions on scan, or clinical or neurologic worsening despite stable disease on the last 2 scans.
3. Patients may have had any number of prior surgeries, radiation and/or chemotherapy regimens as adjuvant, neoadjuvant or palliative therapy for the treatment of their disease
4. Patients must be >/=18 years of age.
5. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2.
6. Patients must have adequate bone marrow function as evidenced by an absolute neutrophil count >/=1,500/microliters and a platelet count >/=100,000/microliter, adequate renal function as evidenced by serum creatinine </=2.0 mg/dL, adequate hepatic function as evidenced by serum total bilirubin </=2.0 mg/dL, AST/serum glutamate oxaloacetate transaminase (SGOT) and ALT/serum glutamate pyruvate transaminase (SGPT) </= 3X the upper limit of normal (ULN).
7. Patients must have recovered and healed from the effects of any prior surgery, must have received prior chemotherapy at least 2 weeks prior to dosing with adequate recovery of white blood cell count (WBC) and platelet counts, and at least 12 weeks must have elapsed from the completion of radiotherapy, unless there are new lesions appearing on imaging within this 12 weeks frame.
8. Women of child-bearing potential (i.e. </= 50 years of age or has had menstrual cycle within the past 12 months, if > 50 years of age. If in doubt, check FSH, LH and estradiol level) must have a negative urine or serum pregnancy test at screening.
9. Sexually active patients must agree to use adequate contraception (abstinence or barrier contraceptives must be used throughout the trial and one month after end of treatment) for the duration of the study .
10. Patients or their legal representative must be able to read, understand and sign an informed consent form (ICF).
11. TPI 287 may interfere with coumadin dosing and patients who are taking this combination will require monitoring of their PT, PTT and international normalized ratio (INR).

Exclusion Criteria:

1. Patients who are receiving concurrent enzyme-inducing anti-epileptic drugs (EIAEDs) (e.g., carbamazepine, oxcarbazepine, phenytoin, fosphenytoin, phenobarbital and primidone) or who received EIAEDs within 2 weeks prior to the first dose of study drug.
2. Patients with uncontrolled intracranial hypertension syndrome (defined as: persistence of headache, transient visual obscurations, and/or diplopia despite optimal clinical management) or uncontrolled seizure activity (i.e. recorded despite optimal medical management).
3. Patients who are not on a stable or decreasing steroid dose for the previous week prior to the first dose of study enrollment
4. Patients who are taking bevacizumab or have taken bevacizumab within the past 2 weeks for treatment of their brain metastases
5. Patients with an active infection (i.e., clinical signs or symptoms, including, but not limited to: bleeding/pustulant skin infections; productive cough associated with fever) on antibiotics or with a fever >/=38.5°C within 3 days prior to registration (i.e. date when the patient signs the consent and/or the patient is registered in CORE).
6. Patients with New York Heart Association (NYHA) Class 3 or 4 congestive heart failure.
7. Patients with known HIV or Hepatitis B or C
8. Patients who are pregnant or lactating or not practicing adequate contraception
9. Patients with any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with the patient's ability to sign the ICF or his/her ability to cooperate and participate in the study, or to interfere with the interpretation of the results.
10. Patients who are receiving concomitant systemic therapy for breast cancer.
11. Patients with leptomeningeal disease (LMD) or with a history of LMD will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-08-16 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2017-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nuhad K. Ibrahim, MD,BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.utmdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Metastatic breast cancer any receptors status with brain metastasis
Groups:
- TPI 287: TPI 287 administered at 160 mg/m2 by vein on Day 1 and repeated every three weeks. Day 1 of each subsequent cycle is equivalent of day 22 of the previous cycle; pre TPI 287: Dexamethasone 6 mg by mouth at 12 hours and 6 hours prior to treatment. As alternative and based on the treating physician discretion, Dexamethasone 10 mgby vein may be given 30-60 minutes prior to treatment with TPI 287, Benadryl 12.5-25 mg IV push over 30-60 minutes, and Ranitidine 1mg/kg IV over 30-60 minutes.
  TPI 287: Starting dose Phase I: 160 mg/m2 by vein over 60 minutes on Days 1, 8, and 15 of every 28 day cycle.
  Starting Dose Phase II: Maximum tolerated dose from Phase I.
  Dexamethasone: 6 mg by mouth at 12 hours and 6 hours prior to treatment. As alternative and based on the treating physician discretion, dexamethasone 10 mg by vein may be given 30-60 minutes prior to treatment with TPI 287.
  Benadryl: 12.5-25 mg intravenous (IV) push 30-60 minutes prior
  Ranitidine: As H2 blocker 1mg/kg IV
Period: Overall Study
Arm/Group | TPI 287
Started | 24
Completed | 21
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: All patient's enrolled in the study were analyzed (Intention To Treat)
Groups:
- Phase 1/2: TPI 287 administered at 160 mg/m2 by vein on Day 1 and repeated every three weeks. Day 1 of each subsequent cycle is equivalent to day 22 of the previous cycle; pre TPI 287: Dexamethasone 6 mg by mouth at 12 hours and 6 hours prior to treatment. As alternative and based on the treating physician discretion, Dexamethasone 10 mg by vein may be given 30-60 minutes prior to treatment with TPI 287, Benadryl 12.5-25 mg IV push over 30-60 minutes, and Ranitidine 1mg/kg IV over 30-60 minutes.
Arm/Group | Phase 1/2
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 45 [28 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR."
Time Frame: 8-24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- TPI 287: TPI 287 administered at 160 mg/m2 by vein on Day 1 and repeated every three weeks. Day 1 of each subsequent cycle is equivalent of day 22 of the previous cycle; pre TPI 287: Dexamethasone 6 mg by mouth at 12 hours and 6 hours prior to treatment. As alternative and based on the treating physician discretion, Dexamethasone 10 mg by vein may be given 30-60 minutes prior to treatment with TPI 287, Benadryl 12.5-25 mg IV push over 30-60 minutes, and Ranitidine 1mg/kg IV over 30-60 minutes.
Arm/Group | TPI 287
Number analyzed (Participants) | 21
Participants | 21

ADVERSE EVENTS:
Time Frame: Collected every 28 days with an average of up to a year.
Arm/Group | TPI 287
All-Cause Mortality (participants affected / at risk) | 1/21
Serious Adverse Events (participants affected / at risk) | 6/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TPI 287 (N=21)
Dizziness (Nervous system disorders) | 3
Syncope (Nervous system disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Fracture (Musculoskeletal and connective tissue disorders) | 1
Hypertension (Cardiac disorders) | 3
Edema (Cardiac disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TPI 287 (N=21)
Alopecia (Skin and subcutaneous tissue disorders) | 3 — Grade 2
Anemia (Blood and lymphatic system disorders) | 3 — Grade 2
Anemia (Blood and lymphatic system disorders) | 1 — Grade 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 — Grade 2
Decreased ANC (Blood and lymphatic system disorders) | 7 — Grade 2
Decreased ANC (Blood and lymphatic system disorders) | 2 — Grade 3
Decreased Lymphocytes (Blood and lymphatic system disorders) | 6 — Grade 2
Decreased Lymphocytes (Blood and lymphatic system disorders) | 2 — Grade 3
Decreased WBC (Blood and lymphatic system disorders) | 3 — Grade 2
Dizziness (Nervous system disorders) | 1 — Grade 2
Dizziness (Nervous system disorders) | 1 — Grade 3
Dysphagia (Nervous system disorders) | 1 — Grade 2
Dysphagia (Nervous system disorders) | 2 — Grade 3
Dyspnea (Nervous system disorders) | 1 — Grade 2
Increased alk phos (Blood and lymphatic system disorders) | 1 — Grade 2
increased AST (Blood and lymphatic system disorders) | 1 — Grade 2
Edema limbs (Cardiac disorders) | 1 — Grade 2
Fatigue (Metabolism and nutrition disorders) | 10 — Grade 2
Fatigue (Metabolism and nutrition disorders) | 5 — Grade 3
Fever (Immune system disorders) | 1 — Grade 2
Fracture (Musculoskeletal and connective tissue disorders) | 2 — Grade 3
Hand foot syndrone (Immune system disorders) | 3 — Grade 2
Headache (Nervous system disorders) | 1 — Grade 3
Hyperglycemia (Endocrine disorders) | 1 — Grade 3
HTN (Cardiac disorders) | 1 — Grade 2
Hypoalbuninemia (Blood and lymphatic system disorders) | 1 — Grade 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 — Grade 2
Infection (Infections and infestations) | 1 — Grade 2
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 2 — Grade 2
Nausea (Gastrointestinal disorders) | 2 — Grade 3
Neuropathy (Nervous system disorders) | 7 — Grade 2
Pain (General disorders) | 5 — Grade 2
Pain (General disorders) | 3 — Grade 3
Seizure (Nervous system disorders) | 1 — Grade 2
Skin tissue disorder (Skin and subcutaneous tissue disorders) | 2 — Grade 2
Syncope (Cardiac disorders) | 1 — Grade 3
Vaginal candidiasis (General disorders) | 1 — Grade 2
Vomiting (Gastrointestinal disorders) | 1 — Grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT01332630/Prot_SAP_000.pdf